CLINICAL TRIAL: NCT01899404
Title: A Pilot Prospective Study of the Utility of Dynamic Contrast-Enhanced Magnetic Resonance Imaging (DCE-MRI), Diffusion Weighted MRI (DWI)and Positron Emission Tomography (PET) Imaging With 18F-Fluorodeoxyglucose (18FDG) in Brachytherapy for Cervix Cancer
Brief Title: MRI FDG PET Imaging Cervix
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Collaborators: Princess Margaret Hospital, Canada (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN REB 12-5221-C
Record Dates: First submitted 2012-10-23; First posted 2013-07-15 (Estimated); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Cervical Cancer Squamous Cell
Keywords: Cervical Cancer; PET Scan for cervix; MRI for cervix
MeSH Terms: conditions — Uterine Cervical Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 18-FDG PET/CT, DWI, DCE-MRI (Experimental)
  Interventions: Biological: 18-FDG PET/CT, DWI, DCE-MRI

INTERVENTIONS:
Biological: 18-FDG PET/CT, DWI, DCE-MRI — All patients on this study will receive a Diffuse Weighted MRI and Dynamic Contrast Enhancing MRI during the routine MRI session on the day of brachytherapy (additional 10 minutes), and a FDG PET/CT scanning session on the day of brachytherapy.

SUMMARY:
The standard treatment for cervix cancer at Princess Margaret Hospital is external radiation with chemotherapy followed by internal radiation, called brachytherapy. Currently, brachytherapy treatment is planned on a type of Magnetic Resonance Imaging (MRI) called T2-weighted (T2W) MRI.

The main purpose of this study is to determine whether the following imaging tests can visualize the tumor better for planning the brachytherapy treatment:

1. special types of MRI called diffusion weighted MRI (DWI) and dynamic-contrast enhanced MRI (DCE-MRI); and
2. an x-ray test called positron emission test (PET) performed with a sugar dye called FDG. MRI-guided brachytherapy is resource-intensive and not widely available.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Histologic diagnosis of squamous cell carcinoma, adenocarcinoma or adenosquamous carcinoma of the cervix
3. FIGO Stage IB - IVA
4. Intention to treat using radiotherapy with or without concurrent cisplatin chemotherapy according to the current treatment policies of the PMH Gynecology Group
5. Intention to treat with MR-guided brachytherapy as part of standard radiotherapy according to the current treatment policies of the PMH Gynecology Group
6. No cytotoxic anti-cancer therapy for cervix cancer prior to study entry
7. A negative urine or serum pregnancy test within the two week interval immediately prior to the first PET-CT imaging, in women of child-bearing age
8. Ability to provide written informed consent to participate in the study

Exclusion Criteria:

1. Prior complete or partial hysterectomy
2. Carcinoma of the cervical stump
3. Inability to lie supine for more than 30 minutes
4. Insulin-dependent diabetes mellitus
5. Impaired kidney function with glomerular filtration rate < 30
6. Previous anaphylactic reaction to gadolinium or other contraindications to MR.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-10-03 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Target delineation in brachytherapy using standard T2-weighted MRI versus DCE-MRI, DWI and FDG-PET/CT imaging: gross tumor volume and high-risk clinical target volume in patients with cervical cancer | 2 years
Target delineation using standard MRI acquired during the last week of EBRT fused to planning CT versus full MRI-guided brachytherapy. | 2 years
  This objective will evaluate the potential for translation of this technique to centres with limited MRI access.

SECONDARY OUTCOMES:
Follow-up imaging (MRI and 18FDG PET) versus the imaging done at the time of brachytherapy | 2 years
Imaging techniques for visualizing the brachytherapy applicator. | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kathy Han, MD, Principal Investigator — University Health Network, The Princess Margaret
Locations (1):
- University Health Network, The Princess Margaret, Toronto, Ontario, Canada